CLINICAL TRIAL: NCT04526080
Title: A Randomized Phase II Study Of Intrabucally Administered Electromagnetic Fields Versus Placebo as Third-line Therapy For Patients With Advanced Hepatocellular Carcinoma
Brief Title: Intrabucally Administered Electromagnetic Fields Versus Placebo as Third-line Therapy For Patients With Advanced Hepatocellular Carcinoma
Acronym: TheraBionics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This application needs further attention in terms of FDA approval and will be reassigned under a different trial number later.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00068320; WFBCCC 55320 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TheraBionic Arm (Experimental): Self-administered from the device that delivers low levels of radiofrequency electromagnetic fields into the body with a spoon-shaped antenna placed in the mouth.
  Interventions: Device: TheraBionic Device
- Placebo Arm (Placebo Comparator): Placebo device that looks and sounds like the active device.
  Interventions: Device: Placebo Device

INTERVENTIONS:
Device: TheraBionic Device — Amplitude-modulated electromagnetic fields will be self-administered and given continuously to patients in three courses of 60-minute treatments per day, administered in the morning, at noon and in the evening at the patient's home, with the exception of the first 60-minute treatment, which will be delivered at the research site. Each 6-week treatment period will be considered a cycle of treatment. For subjects who are randomized to the active arm, the device will be programmed with hepatocellular carcinoma-specific modulation frequencies and will be activated for more than 200 one-hour treatment sessions.
  Arms: TheraBionic Arm
Device: Placebo Device — Subjects who are randomized to receive placebo, will receive the same instructions and a similar device. The placebo device will look and sound the same as the active device, but will not deliver the modulation frequencies. For subjects randomized to the placebo arm, the device will not emit any hepatocellular carcinoma-modulation frequencies and will be activated for more than 200 one-hour treatment sessions.
  Arms: Placebo Arm

SUMMARY:
The primary goal of this study is to gather efficacy data concerning overall survival with electromagnetic field when compared to a placebo amplitude-modulated radiofrequency electromagnetic field device in subjects who have failed or are intolerant to at least two previous systemic therapies

DETAILED DESCRIPTION:
Primary Objective: To estimate overall survival.

Secondary Objectives

* To estimate progression-free survival.
* To evaluate safety and tolerability in this patient population.
* To evaluate the effect on levels of alpha-fetoprotein.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven hepatocellular carcinoma that is locally advanced or metastatic
* Patients must have measurable disease.
* Failure or intolerance to prior treatments with at least two different approved or experimental systemic therapies including sorafenib, lenvatinib, regorafenib, cabozantinib, ramucirumab, nivolumab, nivolumab plus ipilumab, atezolizumab and bevacizumab, or any approved or experimental first line and/or second line therapy that did not include the TheraBionic device (defined as documented radiological progression according to the radiology charter). Randomization needs to be performed within 10 weeks after the last systemic treatment
* Measurable disease according to mRECIST for hepatocellular carcinoma.
* At least one target lesion should not have previously received any local therapy, such as surgery, radiation therapy, hepatic arterial embolization, TACE, hepatic arterial infusion, radio-frequency ablation, percutaneous ethanol injection or cryoablation, unless it has subsequently progressed by 20% or more according to mRECIST for hepatocellular carcinoma.
* Patients with Child's Pugh A or B (at time of enrollment) as defined by the parameters contained in the Child Pugh Calculator.-Subjects with Child's Pugh score of B8-B9 may be included if they have: Albumin > 2.8 mg/l AND Total Bilirubin < 3.0mg/l, Performance status ECOG 0-2.
* Patient must not have curative treatment options, including surgery or radiofrequency ablation, available as assessed by their physician.
* Any extra-hepatic metastases, including treated CNS metastases but patients cannot have leptomeningeal disease.
* At least 4 weeks must have elapsed since administration of any anti-cancer treatment.
* Other anti-cancer treatments are not permitted during this study
* Patients must be more than 18 years old and must be able to understand and sign an informed consent.
* Patient must agree to be followed up according to the study protocol.

Exclusion Criteria:

* Known leptomeningeal disease.
* Fibro lamellar hepatocellular carcinoma.
* Patients with any of the following history within the 12 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.
* Pregnant or breastfeeding women
* Has received treatment for other carcinomas within the last three years except for cured non-melanoma skin cancer, low-risk prostate cancer, T1/T2 glottic cancer, stage 0 or stage I breast cancer, non-invasive bladder cancer, or treated in-situ cervical cancer).
* Patients receiving calcium channel blockers and any agent blocking L-type of T-type Voltage Gated Calcium Channels, e.g. amlodipine, nifedipine, ethosuximide, ascorbic acid (vitamin C), etc. are not allowed in the study unless their medical treatment is modified to exclude calcium channel blockers prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 6 months
  Overall survival will be assessed on an intention to treat basis using a 2-sided log rank test to compare hazard rates between groups. Kaplan-Meier survival curves will also be generated and median survival and corresponding 95% confidence intervals will be estimated for each group.

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 2 years
  Progression free survival (PFS) will be compared between groups using a 2-sided log rank test. Kaplan-Meier survival curves for PFS will also be generated and median progression free survival and corresponding 95% confidence intervals will be estimated for each group.
Proportion of Patients Progression Free After 12 weeks | 12 weeks, 4 months and 6 months
  Proportion of patients who are progression free after 12 weeks (after 2nd 6-week visit) and compare this between groups using a Fisher's exact test. In addition, the corresponding 95% Clopper Pearson exact confidence intervals will be calculated for the 4 month and 6 month progression free survival rates
Number of Adverse Events | Up to 28 days after last study treatment administration
  Type, incidence, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 5.0), timing, seriousness, and relatedness of adverse events and laboratory abnormalities. adverse events will be compared for each CTL type between the two groups using the Fisher's exact test (two-sided) at level 0.05. These comparisons will be made to compare events of grade greater than or equal to 3 between each group.
Changes in Alfa-Fetoprotein Levels | 6 months
  Average alfa-fetoprotein levels will be examined over time, and these changes in alfa-fetoprotein rates after 6 months will be examined for each response category (complete response, partial response, stable disease, progressive disease) and tested using a 1-way ANOVA to see if the change in alfa-fetoprotein level differs by response category.
Response Rates | 6 months
  Response rates we will estimate the proportion of patients who respond and the corresponding 95% Clopper Pearson exact confidence intervals. Patients who are removed from study before the 6-month time point will be considered to not have disease control at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: William Blackstock, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No